CLINICAL TRIAL: NCT00166582
Title: Parent-Youth Teamwork in Pediatric Asthma Management
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R03HD039767 (NIH)
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2007-07-02 (Estimated); Status verified 2005-11

CONDITIONS: Asthma
Keywords: pediatric asthma, medication adherence, adolescents
MeSH Terms: conditions — Asthma; Medication Adherence

INTERVENTIONS:
Device: electronic medication monitoring system
Behavioral: parent-adolescent communication and problem-solving skills

SUMMARY:
The purpose of this research study is to examine the effectiveness of a parent-youth teamwork treatment and an asthma education treatment in helping children use their asthma medicines correctly. We also want to learn about how these treatments affect parental involvement in asthma care, parent and youth relationships, and children's health care.

DETAILED DESCRIPTION:
Noncompliance with medication is a prevalent problem for pediatric asthma patients, particularly for pre-adolescents and adolescents. Families reportedly struggle with the transition of expecting adolescents to assume more independence and responsibility in asthma management. Parent-child collaborative management of pediatric chronic illness regimens has been related to better adherence to medical regimens and improved health outcome. This study has four aims. The first aim is to investigate the effectiveness of a low-intensity, behavioral intervention aimed at promoting parental involvement in children's asthma management, particularly in improving medication adherence. The second aim is to examine how the role of parental involvement changes across time and participation in a 5-month study. A third aim is to determine whether parent-adolescent conflict is changed by the intervention. The fourth aim is to evaluate whether participation in the treatment program is associated with improved health status (e.g., improved pulmonary function test results).

Established asthma patients (ages 9-15) will be randomly assigned to one of three groups: Treatment Intervention (TI), Asthma Education (AE), and Standard Care (SC). The TI and AE groups will receive four 30-minute treatment sessions every two weeks. The TI intervention will consist of strategies aimed at promoting parent-youth management in asthma management. The AE group will receive structured reviews of asthma educational materials typically given to asthma patients. SC participants will have no contact with researchers beyond that necessary to gather data. Data will be collected from all participants every two weeks for the first 8-weeks of study involvement and also about 3-months after the final treatment session. Outcome data will include objective measures of medication adherence, parental involvement in asthma, and health outcome.

ELIGIBILITY:
Inclusion Criteria:

* patient has been diagnosed with asthma for at least 6 months
* patient can be managed appropriately on study medications as determined by the attending physician

Exclusion Criteria:

* patient shows evidence of neurological or significant cognitive impairment

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60
Dates: Start 2002-04; Study Completion 2005-09

PRIMARY OUTCOMES:
medication adherence, parental involvement , perceived parent-adolescent conflict, associated health outcome

CONTACTS AND LOCATIONS:
Overall Officials: Christina D Adams, PhD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (2):
- United States (2):
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - West Virginia Univeristy, Morgantown, West Virginia

REFERENCES:
- [Derived] Duncan CL, Hogan MB, Tien KJ, Graves MM, Chorney JM, Zettler MD, Koven L, Wilson NW, Dinakar C, Portnoy J. Efficacy of a parent-youth teamwork intervention to promote adherence in pediatric asthma. J Pediatr Psychol. 2013 Jul;38(6):617-28. doi: 10.1093/jpepsy/jss123. Epub 2012 Dec 17. PMID 23248342